CLINICAL TRIAL: NCT04935320
Title: Phase 1, Randomised, Open-label, 3-period Crossover, Single Dose Study in Healthy Subjects, to Assess Relative Bioavailability From an Oral Capsule of HTL0016878 Citrate Salt Versus an Oral Solution of HTL0016878 Hydrochloride Salt
Brief Title: Comparison of Blood Levels of HTL0016878 From an Oral Capsule and an Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HTL0016878-102; 18-018 (Other: Hammersmith Medicines Research Ltd); 2018-003685-14 (EudraCT Number)
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
Keywords: Relative Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Solution Fasted (Experimental): HTL0016878.HCl 10 mg, single dose, oral solution, fasted
  Interventions: Drug: HTL0016878.HCl Solution 10 mg
- Oral Capsule Fasted (Experimental): HTL0016878.citrate 10 mg, single dose, oral capsule, fasted
  Interventions: Drug: HTL0016878.Citrate Capsule 10 mg
- Oral Capsule Fed (Experimental): HTL0016878.citrate 10 mg, single dose, oral capsule, fed
  Interventions: Drug: HTL0016878.Citrate Capsule 10 mg

INTERVENTIONS:
Drug: HTL0016878.HCl Solution 10 mg — Oral solution fasted
  Arms: Oral Solution Fasted
Drug: HTL0016878.Citrate Capsule 10 mg — Oral capsule fed or fasted
  Arms: Oral Capsule Fasted; Oral Capsule Fed

SUMMARY:
This is a randomised, open-label, 3-period, crossover single dose study to assess the relative bioavailability of two formulations of HTL0016878: an oral solution of HCl salt form (the reference product) and an oral capsule containing citrate salt (the test product); and of the effect of food on the pharmacokinetics of the capsule formulation.

DETAILED DESCRIPTION:
Fifteen healthy male or female subjects will be enrolled. Each subject will have 3 study sessions and receive a single oral dose of 10 mg HTL0016878 on Day 1 of each study session. Subjects will receive the HTL0016878.HCl oral solution in the fasted state in 1 session, and the HTL0016878.citrate capsule, in the fasted state and after a high-fat meal, respectively, in the other 2 sessions. Each subject will be randomised to 1 of 3 treatment sequences (5 subjects to each sequence). There will be a washout of at least 10 days between doses. Subjects will be screened within 35 days before their first dose of HTL0016878. In each study session, subjects will be resident on the ward from the day before dosing (Day -1) until completion of procedures 72 h after their dose (Day 4). Subjects will return for a follow up visit 10-13 days after their final dose of trial medication.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or females, aged 18-50 years
2. Female subjects must agree to use highly effective contraception
3. Weigh 60 kg or more, with a BMI in the range 18.0-30.0 kg/m2
4. Sufficient intelligence to understand the nature of the trial
5. Willingness to give written consent to participate
6. Agree to use the contraception requirements of the trial
7. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication
8. Willingness to give written consent to have data entered into The Overvolunteering Prevention System

Exclusion Criteria:

1. Woman who is pregnant or lactating
2. Clinically relevant abnormal history, physical findings, ECG, or laboratory values
3. Presence or history of acute or chronic illness, or mental health problem
4. Impaired neurological, endocrine, thyroid, cardiovascular, respiratory, gastrointestinal, hepatic or renal function, diabetes mellitus, coronary heart disease, or history of any psychiatric disorder or psychotic mental illness
5. Cancer during the 5 years before screening
6. Supine blood pressure and heart rate outside the ranges: 90-140 mm Hg systolic and 50-90 mm Hg diastolic blood pressure; heart rate 45-80 beats/min
7. Supine QT interval (QTcF) outside the ranges 300-450 msec (men) and 300-470 msec (women)
8. Personal or family history of long QT syndrome or family sudden death
9. Positive test for hepatitis B, hepatitis C or HIV
10. Aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase or total bilirubin levels > 1.5 times the upper limit of normal
11. Creatinine clearance < 80 mL/min/1.73 m2
12. Presence or history of drug or alcohol abuse in the past 5 years; or regular intake of more than 21 units of alcohol weekly (for men) or 14 units of alcohol weekly (for women); or use of cigarettes, tobacco and/or nicotine-containing products during the 3 months before dosing
13. Evidence of drug abuse or positive alcohol or cotinine test results
14. Positive pregnancy test
15. Habitual and heavy consumption of caffeinated beverages
16. Use of a prescription or over-the-counter medicine, any herbal remedy, or nutritional supplement
17. Receipt of a vaccine against COVID-19 in the 14 days before dosing
18. Received live attenuated vaccination within 6 weeks prior to Screening
19. History of severe allergies
20. Use of any drugs that are inhibitors of CYP2D6
21. Poor metaboliser of CYP2D6
22. History of epilepsy or seizures
23. Any disease associated with cognitive impairment and/or psychosis
24. Suicidal thoughts or ideation, or insomnia
25. Any history of mental illness (including anxiety, depression), which required medical intervention
26. Presence or history of severe adverse reaction to any drug
27. Surgery or medical condition that might affect absorption of medicines
28. Receipt of an investigational product as part of another clinical trial within the 3 months before dosing in this study
29. Receipt of HTL0016878 in a previous clinical trial
30. Loss of more than 400 mL blood during the 3 months before dosing
31. Unwilling to eat a high-fat breakfast
32. Possibility that the volunteer will not cooperate with the requirements of the protocol
33. Objection by GP to volunteer entering trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Concentration of HTL0016878 in plasma Cmax | 0-72 hours
  Pharmacokinetics
Concentration of HTL0016878 in plasma AUC | 0-72 hours
  Pharmacokinetics

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | Baseline up to 13 days post-dose
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd (HMR), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No